CLINICAL TRIAL: NCT04901884
Title: Exploratory Evaluation of Simultaneous Cardiac PET/MR, Metabolomic Markers and Circulating DNA as Possible Prognostic Markers in Identifying Patients Developing Transient or Permanent Cardiopulmonary Dysfunctions After Radiotherapy
Brief Title: PET/MR Pre- and Post Radiotherapy for Cardiopulmonary Dysfunction Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-5879
Record Dates: First submitted 2021-03-17; First posted 2021-05-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Biopsy or otherwise clinically proven thoracic malignant mass which is intended to be treated with radio(chemo)therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm / exploratory study (Experimental): Injection of 18F-FDG.The 18F-FDG cardiac PET-MR scanning visit will take up to 1.5 hours.
  Interventions: Drug: PET/MR with 18F-FDG

INTERVENTIONS:
Drug: PET/MR with 18F-FDG — (18F) Fluorodeoxyglucose (FDG) will be administered by intravenous injection at a dose of 4-5 MBq/kg.

SUMMARY:
Radiotherapy (RT) is a well-known and established therapy or adjuvant therapy for the treatment of thoracic cancer It uses a high energy radiation from x-rays, gamma rays and other charged particles that assist in damaging the cancer DNA.

PET/MR as imaging biomarkers for cardiopulmonary dysfunction with a focus on Pulmonary hypertension (PH).

Despite the measures taken to reduce the total radiation dose and to limit the radiation to normal tissues, there is evidence of transient or permanent radiotherapy induced myocardial and pulmonary dysfunction leading to PH in patients who receive radiotherapy above a certain threshold of received dose.

To be able to Demonstrate correlation of combined PET/MR and plasma metabolomics markers in patients at risk of developing cardiopulmonary disfunction after RT.

DETAILED DESCRIPTION:
RT is a well-known and established therapy or adjuvant therapy for the treatment of thoracic malignancies (breast cancer, lung cancer, lymphoma and others). It usually uses high energy radiation from x-rays, gamma rays or other charged particles to induce DNA damage in malignant cells. Despite the measures taken to reduce the total radiation dose and to limit the radiation to normal tissues, the signs and symptoms of radiation induced cardiopulmonary dysfunction (RICPD) still persist. However, in the majority of cases, it remains unclear which cardiopulmonary damage is the main /leading cause for the clinical symptoms the patients are experiencing.

Hybrid PET/MRI is a promising technique that allows for truly simultaneous molecular, anatomic and functional imaging of the cardiopulmonary system. The simultaneity is an important aspect in this proposed study since only parameters measured at the same time in PET and MR can be used for an integrated, multimodality parameter for possible detection and prognostication of the different underlying processes of cardiopulmonary dysfunction after RT. Furthermore, certain PET-uptake of the RV have to be corrected for RV mass which is only possible with concomitant anatomical imaging. MR imaging and PET at different time point are not accurately reflective of the underlying pathophysiological pathways and metabolic state at the specific time points pre- and post radiotherapy. To our knowledge, there are no online publications of its use in the diagnosis and prognostication of cardiopulmonary dysfunction after RT and specifically PH.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Biopsy or otherwise clinically proven thoracic malignant mass which is intended to be treated with radio(chemo)therapy
* Intention to treat with radio(chemo)therapy with incidental cardiac irradiation of at least 25Gy.
* A negative urine or serum pregnancy test within the two week interval immediately prior to imaging, in women of child-bearing age.
* Ability to provide written informed consent to participate in the study (for all components of the trial: imaging with cardiac PET/MR, blood sampling for plasma metabolomics and circulating DNA).

Exclusion Criteria:

* Contraindication for MR as per current institutional guidelines.
* Contraindication for Gadolinium injection as per current institutional guidelines.
* Inability to lie supine for at least 45 minutes.
* Any patient who is pregnant or breastfeeding.
* Any patient with known hypersensitivity to 18F-FDG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change of FDG uptake of heart | at 4 weeks prior to radiotherapy, and at 6-10 weeks after completion of radiotherapy
  FDG uptake of the left and right ventricles of heart will be measured and compared in PETMRI scans
Change of FDG uptake of lungs | at 4 weeks prior to radiotherapy, and at 6-10 weeks after completion of radiotherapy
  FDG uptake of left and right ratios within the lungs in PETMRI scans
Change of the heart function | at 4 weeks prior to radiotherapy, and at 6-10 weeks after completion of radiotherapy
  MRI of ventricular volumes in PETMRI scans
Change of the lung perfusion | before radiotherapy and up to 16 weeks after completion of radiotherapy
  Percentage of the perfused/ventilated lung segments will be evaluated and compared pre and post therapy by SPECT scans

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada